CLINICAL TRIAL: NCT05511441
Title: Routine Minimally Invasive Thoracic Surgery Without Aspirin Withdraw Before Surgery
Brief Title: Routine Minimally Invasive Thoracic Surgery Without Aspirin Withdraw
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aspirin ZYP
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Aspirin Sensitivity; Surgery
Keywords: Aspirin; Minimally Invasive Thoracic Surgery; Safety
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery Without Aspirin Withdraw (Experimental): Routine Minimally Invasive Thoracic Surgery Without Aspirin Withdraw
  Interventions: Procedure: Surgery Without Aspirin Withdraw

INTERVENTIONS:
Procedure: Surgery Without Aspirin Withdraw — Routine Minimally Invasive Thoracic Surgery Without Aspirin Withdraw

SUMMARY:
Surgeons are increasingly confronted by patients on long-term low-dose acetylsalicylic acid (ASA). However, the perioperative management of these patients undergo non-cardiac surgery has not yet been clear. This single- arm study was to evaluate the safety of continuous use of ASA in the perioperative period in routine minimally thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients with stage I-IIIa Non-small-cell Lung Cancer underwent radical resection or other benign lung lesions need Minimally Invasive Thoracic Surgery;
2. VATS and robotic surgery are both permitted;
3. cardio-pulmonary function can tolerate surgery.

Exclusion Criteria:

1. cardio-pulmonary function couldn't tolerate surgery;
2. high bleeding risk after the pre- operative evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
bleeding volume | on the surgery day
  bleeding volume during surgery
surgery time | on the surgery day
  total surgery time
postoperative drainage volume | within 7 days after surgery
  chest drainage volume after surgery
postoperative drainage duration | within 7 days after surgery
  chest drainage duration after surgery
postoperative hospitalization time | within 7 days after surgery
  postoperative hospitalization time
postoperative complication rate | within 14 days after surgery
  postoperative complication rate

SECONDARY OUTCOMES:
progression- free survival | within 5 years after surgery
  progression- free survival
overall survival | within 10 years after surgery
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Study Director — The Second Hospital of Shandong University
Locations (1):
- The Second Hospital Of Shandong Univercity, Jinan, Tianqiao, China